CLINICAL TRIAL: NCT06361732
Title: Prevalence of CYP3A5 Polymorphisms in the Donors and ABCB1 Polymorphisms in the Recipients Undergoing Pediatric Liver Transplant and Their Influence on Tacrolimus Levels and Graft Function.
Status: Recruiting | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-liver Transplant-03
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Pediatric Liver Transplant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver Transplant: Liver Transplant
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
It is known that Immunosuppression post-Liver transplant is central to achieving optimal outcomes in liver transplant recipients. It is required to maintain an adequate balance between reducing rejection and toxicities. Mainstay drugs for maintenance therapy are Calcinuerin inhibitors - Tacrolimus versus cyclosporine. Tacrolimus is preferred, as it has less rejection and better graft survival. However, there is risk of renal and metabolic toxicities. Tacrolimus is bound mainly to alpha1-acid-glycoprotein (encoded by the ABCB1gene) expressed on various epithelial and endothelial cells and lymphocytes. Elimination occurs by metabolizing enzymes of cytochrome P450 system, with biliary excretion (95%) of metabolites (majority) with minority through urine (2.4%). Demethylation and hydroxylation of tacrolimus occurs by hepatic and intestinal CYP3A isoforms (CYP3A4 and CYP3A5). Among the factors that play an important role in the pharmacokinetics of tacrolimus, thus affecting the tacrolimus trough levels in the body and in turn influencing the dosing of the drug required to maintain an adequate balance between reducing rejection and toxicities, genetics plays an important role. Increased expression of CYP3A5 causes more metabolism of tacrolimus and hence affecting the tacrolimus concentration/weight-adjusted dose (C/W-D) ratio in the body. The wild type (CYP3A5*3) are slow metabolizers and mutant ones (CYP3A5 *1/*1 and CYP3A5 *1/*3) are fast metabolizers. Fast

metabolizers have a low C/W-D ratio and require higher Tacrolimus dosing and are thus susceptible to renal and metabolic toxicities, EBV viremia and post transplant lymphoproliferative disorder. Polymorphisms in ABCB1 (c.3435C>T) are also known to influence tacrolimus dosage in the first week of transplant (C/D ratio was lower in ABCB1 3435CC in comparison to CT and TT). There is no such data in pediatric liver transplant setting from Indian subcontinent. The aim of the study is to study the prevalence of CYP3A5 polymorphisms in the donors and ABCB1 polymorphisms in the recipients undergoing Paediatric liver transplant and their influence on Tacrolimus levels and graft function.

DETAILED DESCRIPTION:
Aim: To study the prevalence of CYP3A5 polymorphisms in the donors and ABCB1 polymorphisms in the recipients undergoing Paediatric liver transplant and their influence on Tacrolimus levels and graft function.

Primary objective: To compare the time (in days) to achieve transaminases within 1.5 times ULN (60 IU/L) in the pediatric Liver transplant recipients with grafts from slow metabolizer (CYP3A5*3/3 allele) versus fast metabolizer (CYP3A5*1/3 and 1/1 alleles) donors.

Study population: All donors and recipients of Pediatric Liver transplant recipients (0-18 years),from September 2011 till October 2023, follow up atleast 1 for year.

Study design: Retrospective and Prospective. Intervention: None Monitoring and assessment: Monitoring for the Tac C/D levels, graft functions (AST/ALT) , Toxicities of Tacrolimus(neurological,metabolic) and its correlation to the CYP3A5 and ABCB1 polymorphism. This will be as per standard Institutional protocol followed up since the time of start of transplant program.

Polymorphisms in CYP3A5 and ABCB1: Whole blood samples will be collected for donors and recipients in the EDTA vials. DNA extraction will be done as per the standard procedure followed in

the department. Genotype analysis for CYP3A5 (3/3, 3/1 and 1/1) and ABCB1 3435 (CC, CT & TT) alleles will be done by polymerase chain reaction (PCR) amplification and will be detected by restriction fragment length polymorphism (RFLP) analysis.

Statistical Analysis: All the categorical variables will be expressed as frequencies, whereas continuous ones will be expressed as mean+ SD or median (IQR). Chi-square , Fisher's exact test and student's t-test will be applied for assessment of causality. Kaplan-Meier statistics will be done for survival and liver related morbidity besides this an appropriate analysis will be carried out at the time of data analysis like diagnostic test, logistic regression etc. Significance will be mentioned in the form of p-value <0.05.

Adverse effects: No such adverse events are involved in the study

ELIGIBILITY:
Inclusion Criteria:

- All Pediatric Living donor liver Transpalnt Liver transplant recipients (0-18 years of age) from September 2011 till October 2023 with follow-up at least for 1 year.

Exclusion Criteria:

1. Incomplete medical records
2. Non-availability of Donor to check CYP3A5 polymorphism Deceased donor liver transplantation
3. Primary non-function
4. Mortality within 2 weeks of liver transplantation Re-transplantation
5. Children with Hepatitis C infection
6. Multi-visceral or Combined liver-kidney transplantation
7. Hepatic artery thrombosis within 6 months of liver transplantation
8. Biliary complications within 6 months of liver transplantation requiring intervention

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All donors and recipients of Pediatric Liver transplant recipients (0-18 years),from September 2011 till October 2023, follow up atleast 1 for year.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-12-17 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Time (in days) to achieve transaminases within 1.5 times ULN (60 IU/L) in the pediatric Liver transplant recipients with grafts from slow metabolizer (CYP3A5*3/3 allele) versus fast metabolizer (CYP3A5*1/3 and 1/1 alleles) donors. | 1 year

SECONDARY OUTCOMES:
Prevalence of CYP3A5 alleles in the donors of pediatric liver transplant recipients. | Day 0
Influence of donor CYP3A5 alleles (slow versus fast metabolizers) on tacrolimus concentration-weight adjusted dose ratio at 1 week, 4 weeks, 3 months & 6 months and 1 year after liver transplantation. | Day 0
Prevalence of ABCB1 3435 C/T alleles in the recipients of pediatric liver transplant. | Day 0
Influence of recipient ABCB1 3435 C/T on tacrolimus concentration-weight adjusted dose ratio at 1 week, 4 weeks, 3 months and 6 months and 1 year after liver transplantation. | 1 week, 4 weeks, 3 months & 6 months and 1 year.
Comparison of the Number of Rejection episodes 1 year from LT. | 1 year
Comparison of proportion of patients who were withdrawn from Mycophenolate or required addition of Mycophenolate 1 year from LT. | 1 year
Comparison of proportion of patients with renal toxicity 1 year from LT. | 1 year
Comparison of proportion of patients with Neurological toxicity 1 year from LT. | 1 year
Comparison of e-GFRand cystatin-C levels in the two cohorts of pediatric liver transplant recipients with grafts from slow metabolizer (CYP3A5*3/3 allele) versus fast metabolizer (CYP3A5*1/3 and 1/1 alleles) donors. | 6 months and 1 years

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided